CLINICAL TRIAL: NCT00177736
Title: Pharmacodynamic Parameters of Two Different Doses of Cefepime
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: David Paterson, MD, UPMC
Other Study IDs: IRB#0505059
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2007-12-13 (Estimated); Status verified 2007-12

CONDITIONS: Infection; Bacteremia; Pneumonia
Keywords: ventilator associated pneumonia
MeSH Terms: conditions — Infections; Bacteremia; Pneumonia; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Pharmacokinetics is the study of the disposition of drugs in the body, while pharmacodynamics considers the interaction of the drug at the site of infection over time. Mathematical models of antibiotic pharmacodynamics are sometimes used to predict if antibiotic doses are sufficient to treat infection with organisms of different minimal inhibitory concentrations of the antibiotic. Based on these models, there has been speculation that the antibiotic cefepime dosed at one gram every 12 hours, is insufficient to kill all organisms within the "susceptible" range. This study of patients treated with cefepime will involve the collection of blood to determine cefepime concentrations, and determine if those concentrations are effective in killing the bacteria at the site of infection.

DETAILED DESCRIPTION:
This will be a non-interventional study in that the antibiotic and its dose will be chosen by the treating team not the investigators. Patients on cefepime who have ventilator-associated pneumonia or bacteremia will be invited to participate in the study. Blood samples will be taken to determine the pharmacokinetic profile of the drug. Blood cultures will be repeated in patients with bacteremia to determine clearance of infection. A mini-BAL will be repeated in patients with ventilator-associated pneumonia to determine clearance of pneumonia.

ELIGIBILITY:
Inclusion Criteria:

1. Adults of at least 18 years of age or older
2. Culture proven ventilator associated pneumonia (VAP) or bacteremia caused by a cefepime susceptible gram negative pathogen:

   * Bacteremia is defined as at least one positive blood culture
   * VAP is defined by at least 10,000 cfu/ml of an organism from a bronchoalveolar lavage sample
3. Cefepime therapy (1 or 2 grams intravenously [IV] every [q] 8 hours or q 12 hours) initiated as part of standard of care

Exclusion Criteria:

1. Concomitant VAP or bacteremia with a cefepime resistant organism
2. Concomitant therapy with an antimicrobial agent active against gram negative bacilli other than a single dose of aminoglycoside
3. Patients requiring surgical or interventional drainage of purulent collections
4. Pregnant or lactating women
5. Dialysis patients
6. Contraindication to blood sampling
7. Cystic fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2005-09; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L Paterson, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States